CLINICAL TRIAL: NCT01852461
Title: Perfusion Index Variability in Preterm Infants Treated With Two Different Natural Surfactants for Respiratory Distress Syndrome
Brief Title: Perfusion Index Variability in Respiratory Distress Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Sami Ulus Children's Hospital (Other)
Responsible Party: Principal Investigator, Dilek Dilli, Assos Prof, Dr. Sami Ulus Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 685.114A; Surfactant trial (Other: SamiUlusCH)
Record Dates: First submitted 2013-05-07; First posted 2013-05-13 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Poor Peripheral Perfusion
Keywords: natural surfactants; perfusion index
MeSH Terms: interventions — beractant; poractant alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beractant (Active Comparator): Beractant;bovine lung extract; both initial and subsequent dosing is 100 mg/kg (4 mL/kg), which may be given every 6 hours up to four total doses
  Interventions: Drug: Beractant
- Poractant alfa (Active Comparator): Poractant alfa; porcine lung extract; initial dosing is 200 mg/kg (2.5 mL/kg) and repeated dosing is given at 100 mg/kg (1.25 mL/kg) every 12 hours, up to maximum of two additional doses when indicated
  Interventions: Drug: Poractant alfa

INTERVENTIONS:
Drug: Beractant — Beractant;both initial and subsequent dosing is 100 mg/kg (4 mL/kg), which may be given every 6 hours up to four total doses
  Other Names: Beractant (Survanta)
  Arms: Beractant
Drug: Poractant alfa — porcine lung extract, initial dosing is 200 mg/kg (2.5 mL/kg) and repeated dosing is given at 100 mg/kg (1.25 mL/kg) every 12 hours, up to maximum of two additional doses when indicated
  Other Names: Poractant alfa (curosurf)
  Arms: Poractant alfa

SUMMARY:
Perfusion index may vary according to type of surfactant during the treatment of respiratory distress syndrome.

DETAILED DESCRIPTION:
Peripheral tissues of preterm infants are very sensitive for hypoperfusion, but there are rare data in the literature for peripheral perfusion after surfactant treatment. In this study the investigators aimed to compare the perfusion index (PI) variability in premature infants with respiratory distress (RDS) following instillation of one of two different natural surfactant preparations.

ELIGIBILITY:
Inclusion Criteria:

* premature infants < 32 weeks of gestational age

Exclusion Criteria:

* congenital malformation
* Apgar scores <3 at 5 min

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
perfusion index | 1 week
  PI and oxygen saturation (SpO2) were measured by "Masimo Rainbow SET Radical-7 pulse oximeter" before and after surfactant. The effects of the two treatment regimens on PI, oxygenation and clinical outcome were compared.

SECONDARY OUTCOMES:
Duration of mechanical ventilation | 4 weeks
  The effects of the two treatment regimens on duration of mechanical ventilation were compared

OTHER OUTCOMES:
Mortality | 4 weeks
  The effects of the two treatment regimens on mortality were compared

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Dilli, Assoc Prof, Study Director — Sami Ulus CH